CLINICAL TRIAL: NCT06279767
Title: Efficacy and Safety of TMZ Plus 6-MP in the Patients With Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-557
Record Dates: First submitted 2024-01-31; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma; Cancer; Temozolomide
Keywords: Glioblastoma; Cancer; Temozolomide; 6-mercaptopurine
MeSH Terms: conditions — Glioblastoma; Neoplasms | interventions — Mercaptopurine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with a combination of 6-mercaptopurine and temozolomide (Experimental)
  Interventions: Drug: 6-mercaptopurine

INTERVENTIONS:
Drug: 6-mercaptopurine — 6-mercaptopurine (6-MP) is a crucial drug in the maintenance phase of acute lymphoblastic leukemia treatment.

SUMMARY:
Glioblastoma, the most prevalent malignant tumor in the central nervous system, is characterized by high invasiveness and a propensity to recur, contributing to a relatively elevated mortality rate. Patients diagnosed with high-grade glioblastomas typically experience a median survival period of less than 14 months. Presently, the standard treatment for glioblastoma involves surgical resection combined with postoperative radiotherapy and chemotherapy, with postoperative chemotherapy playing a pivotal role in enhancing patient prognosis. Temozolomide (TMZ), a cutting-edge oral alkylating agent known for its advantageous properties, including easy traversal of the blood-brain barrier, induces DNA alkylation in tumor cells, fostering apoptosis. Currently, it serves as a frontline medication for postoperative chemotherapy in glioblastoma. However, clinical resistance to TMZ chemotherapy significantly hampers its efficacy in later stages. We have recently discovered and validated that 5-aminoimidazole-4-carboxamide (AICA), derived from TMZ, can transform into 5-aminoimidazole-4-carboxamide ribonucleotide-5-phosphate (AICAR) in GBM cells. Hypoxanthine phosphoribosyltransferase 1 (HPRT1) has been identified as the catalyst for the AICA reaction, generating AICAR. AICAR acts as an endogenous activator of AMP-activated protein kinase (AMPK), fostering chemoresistance in glioblastoma through the activation of the AMPK signaling pathway. 6-mercaptopurine (6-MP) competes effectively to inhibit HPRT1 activity, thereby impeding TMZ-induced AMPK activation and significantly heightening glioblastoma cell sensitivity to TMZ. In this project, we propose an innovative strategy involving the combination of 6-MP with TMZ for the treatment of glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65, no gender restrictions.
2. Histologically confirmed glioblastoma as the primary tumor after surgery.
3. Patients with recurrent glioblastoma confirmed by MRI after standard treatment (surgery, Stupp regimen) failure, supported by RANO criteria evaluation.
4. At least one measurable intracranial tumor lesion according to RANO criteria.
5. No prior treatment with 6-mercaptopurine or similar drugs.
6. General condition assessed by Karnofsky Performance Status (KPS) score ≥ 60.
7. Normal bone marrow function: white blood cell count ≥ 3.5 × 10^9/L, neutrophil count ≥ 2.0 × 10^9/L, hemoglobin count ≥ 90 g/L, platelet count ≥ 80 × 10^9/L.
8. Normal organ functions such as heart and lung, and no severe internal diseases.
9. Willing to sign an informed consent form, good compliance, able to attend regular follow-ups, and voluntarily agree to comply with the study protocol.

Exclusion Criteria:

1. Participants who do not consent.
2. Vulnerable populations such as pregnant women, children, and adolescents.
3. No history of or concurrent malignancy within the past 5 years.
4. Abnormal liver function (total bilirubin > 1.5 times the upper limit of normal, ALT/AST > 2 times the upper limit of normal).
5. Impaired kidney function (serum creatinine > 1.5 times the upper limit of normal).
6. Presence of organic heart disease leading to clinical symptoms or cardiac dysfunction (NYHA ≥ Grade 2).
7. Factors significantly affecting oral drug absorption, such as difficulty swallowing, intestinal obstruction, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 12 months
  Progression-free survival (PFS), defined as the time from treatment to progression or death, whichever occurs first

SECONDARY OUTCOMES:
OS | 12 months
  Overall survival (OS), defined as the time from treatment to death
Safety evaluation | 12 months
  Adverse events were assessed according to NCI CTCAE (version 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Yongping You, PhD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Department of Neurosurgery of The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China